CLINICAL TRIAL: NCT02112383
Title: Group Versus Internet-based Cognitive Behavior Therapy for Procrastination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-KI-STUDENT
Record Dates: First submitted 2014-04-06; First posted 2014-04-11 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Procrastination
Keywords: Procrastination; Cognitive behavior therapy; Internet interventions; Group intervention; Students; Randomized controlled trial

ARMS (2):
- Internet-based cognitive behavior therapy (Experimental)
  Interventions: Behavioral: Internet-based cognitive behavior therapy
- Cognitive behavior group therapy (Experimental)
  Interventions: Behavioral: Cognitive behavior group therapy

INTERVENTIONS:
Behavioral: Cognitive behavior group therapy — For participants in the group intervention condition, the modules from a self-help treatment for procrastination will be delivered at four consecutive three-hour sessions at the Student Health Centre at Karolinska Institutet, with approximately two modules given at each session. The sessions will be spaced two weeks apart, during which participants are instructed to complete assignments related to the modules that were in focus of the previous session, e.g., goal-setting, time management, and behavioral experiments, which they are advised to present and discuss with the other participants.
  Arms: Cognitive behavior group therapy
Behavioral: Internet-based cognitive behavior therapy — For participants in the Internet-based condition, the modules from a self-help treatment for procrastination will be distributed weekly during the treatment period, with one module given each week, i.e., ten weeks. In comparison to the group condition, participants will not receive a therapist contact or attend any sessions. In addition, the participants are expected to complete both the reading material and the assignments that are included in each module.
  Arms: Internet-based cognitive behavior therapy

SUMMARY:
Procrastination is defined as a voluntarily delay of an intended course of action despite expecting to be worse-off for the delay, and is considered a persistent behavior pattern that can result in major psychological suffering. About one-fifth of the adult population and half of the student population are presumed having substantial difficulties due to recurrent procrastination in their everyday life. However, chronic and severe procrastinators seldom receive adequate care due to preconceptions and the lack of understanding regarding procrastination and the treatment interventions that are assumed beneficial. Cognitive behavior therapy is often deemed treatment of choice, although the evidence supporting its use is scarce, and only one randomized controlled trial has been performed. The primary aim of the current study is therefore to test the efficacy of cognitive behavior therapy delivered as either a group intervention or via the Internet. Participants will consist of students recruited through the Student Health Centre at Karolinska Institutet. A randomized controlled trial with a sample size of 100 participants divided into two conditions will be employed; a ten week Internet-based cognitive behavior therapy intervention, and an eight week group intervention based on cognitive behavior therapy. The current study is believed to result in two important findings. First, different interventions inherent in cognitive behavior therapy are assumed to be helpful for people suffering from problems caused by procrastination. Second, both a group intervention and an Internet-based cognitive behavior therapy intervention are presumed suitable for administering treatment for procrastination, which is considered highly important as the availability of adequate care is limited, particularly among students. The current study will increase the knowledge regarding the efficacy of different treatments of procrastination, as well as enhance the overall comprehension of the difficulties related to dilatory behavior.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in Swedish
* Computer with Internet access and a working email
* Registered as students at one of the affiliated universities of the Student Health Centre at Karolinska Institutet
* Primary difficulties related to chronic and severe procrastination

Exclusion Criteria:

* Severe depression (30 points or more on MADRS-S)
* Acute conditions in need of treatment; suicidal ideation, neuropsychiatric conditions (ADHD, ADD), misuse of alcohol or drugs, bipolar disorder, schizophrenia, and psychosis
* Ongoing psychotherapy
* Ongoing psychotropic medication (unless dose is stable three months prior the entering treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Pure Procrastination Scale (PPS) | 0 weeks and 8 or 10 weeks
  The PPS features twelve items measuring the prevalence of procrastination.
Change from baseline on the Pure Procrastination Scale (PPS) | 0 weeks and 24 weeks
  The PPS features twelve items measuring the prevalence of procrastination.
Change from baseline on the Procrastination Assessment Scale for Students (PASS) | 0 weeks and 8 or 10 weeks
  The PASS features three items measuring difficulties of procrastination within six different domains of study related activities.
Change from baseline on the Procrastination Assessment Scale for Students (PASS) | 0 weeks and 24 weeks
  The PASS features three items measuring difficulties of procrastination within six different domains of study related activities.

SECONDARY OUTCOMES:
Change from baseline on the Montgomery-Åsberg Depression Rating Scale (MADRS-S) | 0 weeks and 8 or 10 weeks
  The MADRS-S is a self-report version of MADRS and features nine items measuring changes in mood, anxiety, sleeping patterns, appetite, concentration, initiative, emotional engagement, pessimism and attitude towards life.
Change from baseline on the Montgomery-Åsberg Depression Rating Scale (MADRS-S) | 0 weeks and 24 weeks
  The MADRS-S is a self-report version of MADRS and features nine items measuring changes in mood, anxiety, sleeping patterns, appetite, concentration, initiative, emotional engagement, pessimism and attitude towards life.
Change from baseline on the Generalized Anxiety Disorder Assessment (GAD-7) | 0 weeks and 8 or 10 weeks
  The GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Change from baseline on the Generalized Anxiety Disorder Assessment (GAD-7) | 0 weeks and 24 weeks
  The GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Change in baseline on the Symptoms Checklist 90 (SCL-90) | 0 weeks and 8 or 10 weeks
  SCL-90 features 90 items evaluating the participant's physical health and mental well-being, and consists of three global domains as well as nine subdomains.
Change in baseline on the Symptoms Checklist 90 (SCL-90) | 0 weeks and 24 weeks
  SCL-90 features 90 items evaluating the participant's physical health and mental well-being, and consists of three global domains as well as nine subdomains.

OTHER OUTCOMES:
Open-ended questions concerning adverse events | 4/5 weeks, 8/10 weeks, six-month follow-up
  The occurrence and characteristics of possible negative effects of treatment will be examined using open-ended questions, i.e., "did you experience any negative effects during treatment", including rating scales assessing the degree to which the adverse event has affected the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, PhD, Principal Investigator — Stockholm University; David Forsström, MSc, Study Director — Stockholm University; Alexander Rozental, MSc, Study Director — Stockholm University
Locations (1):
- The Student Health Centre at Karolinska Institutet., Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rozental, A., Forsström, D., Nilsson, S., Rizzo, A., & Carlbring, P. (2014). Group versus Internet-based cognitive-behavioral therapy for procrastination: Study protocol for a randomized controlled trial. Internet Interventions, 1(2), 84-89. doi: http://dx.doi.org/10.1016/j.invent.2014.05.005
- [Result] Rozental A, Forsstrom D, Lindner P, Nilsson S, Martensson L, Rizzo A, Andersson G, Carlbring P. Treating Procrastination Using Cognitive Behavior Therapy: A Pragmatic Randomized Controlled Trial Comparing Treatment Delivered via the Internet or in Groups. Behav Ther. 2018 Mar;49(2):180-197. doi: 10.1016/j.beth.2017.08.002. Epub 2017 Aug 5. PMID 29530258
- See also: Official recruitment website — http://www.prokrastinera.se